CLINICAL TRIAL: NCT06217952
Title: A Phase 1, Randomized, Placebo-Controlled, Double Blind Single Ascending Dose Study in Healthy Volunteers to Evaluate the Safety, Tolerability, and Pharmacokinetics of SPL84
Brief Title: Safety, Tolerability, and Pharmacokinetics of SPL84 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SpliSense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SPL84-CL-001-P
Record Dates: First submitted 2023-02-07; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPL84 (Active Comparator)
  Interventions: Drug: SPL84
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SPL84 — SPL84 solution for nebulization
  Arms: SPL84
Other: Placebo — Placebo solution for nebulization
  Arms: Placebo

SUMMARY:
This Phase 1 study evaluated the safety, tolerability, and pharmacokinetics of SPL84 single ascending doses (SAD) in healthy volunteers (HV)

ELIGIBILITY:
Key Inclusion Criteria:

* Male adults 18 to 50 years old
* Considered healthy based on medical history, physical examination, 12-lead ECG and clinical laboratory results
* Body Mass Index (BMI) 19.0-30.0 kg/m2
* Subjects who have no difficulties in receiving drugs by inhalation

Key Exclusion Criteria:

* A major surgical procedure or significant traumatic injury within 28 days prior to study intervention administration
* Recent diagnosis of lung disease (< 12 weeks from planned enrollment)
* Any acute illness (e.g. acute infection) within 48 hours prior to the study intervention administration, which is considered of clinical significance by the Investigator.
* Chronic respiratory disease including but not limited to obstructive airway disease such as asthma or chronic obstructive pulmonary disease (COPD); restrictive disease such as idiopathic pulmonary fibrosis (IPF); or pulmonary vascular disease such as pulmonary arterial hypertension (PAH).
* History of adverse reactions during aerosol delivery of any medicinal product.
* Total body weight ≤50 kg at screening.
* Abnormal forced expiratory volume at one second (FEV1) at screening.
* Oxygen saturation ≤95% at screening.
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transferase (GGT), alkaline phosphatase (ALP) and bilirubin (total and direct) above upper limit of normal (ULN) at screening and clinically significant
* Supine systolic blood pressure <90 or >140 mmHg, supine diastolic blood pressure <50 or >90 mmHg, heart rate <45 or >100 beats per minute (bpm), or elevated body temperature (>38ºC) at screening
* Clinically significant ECG abnormalities at screening
* Positive for SARS-CoV-19 at screening or Day -1 (baseline).
* Positive serology tests for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody at screening.
* Positive urine drug, tobacco, and breath alcohol test result at screening or Day -1 (baseline).
* Use of any prescription or over-the-counter (OTC) medications, including vitamins and herbal or dietary supplements within 14 days prior to dosing.
* Subjects who have received any vaccines within 4 weeks prior to study intervention administration.
* History or current drug/alcohol abuse (excluding use of medicinal cannabis for pain management).
* History of smoking or vaping within 180 days (6 months) of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2023-08-06 (Actual); Study Completion 2023-08-06 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of SPL84 as evaluated by number of subjects with at least one treatment-related adverse event (AE) or serious adverse event (SAEs) | Day 1 through Day 31
  Incidence, nature, and severity of AEs and SAEs
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal heart rate | Day 1 through Day 31
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal respiratory rate | Day 1 through Day 31
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal systolic and diastolic blood pressure | Day 1 through Day 31
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal oximetry | Day 1 through Day 31
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal temperature | Day 1 through Day 31
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal hematology lab test results | Day 1 through Day 31
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal biochemistry lab test results | Day 1 through Day 31
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal urinalysis lab test results | Day 1 through Day 31
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal electrocardiogram (ECG) parameters | Day 1 through Day 31
  using an ECG machine that automatically calculates heart rate and measure PR, QRS, QT, and QTc intervals
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal physical examination findings | Day 1 through Day 31
  Complete physical examinations include general appearance, head, ears, eyes, nose, throat, dentition, thyroid, chest (heart, lungs), abdomen, skin, neurological, extremities, back, neck, musculoskeletal, and lymph nodes.
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal Pulmonary function tests results | Day 1 through Day 31
  Pulmonary function tests will be performed according to the ATS/ERS and FEV1, FVC, and FEF25-75 will be measured

SECONDARY OUTCOMES:
Characterization of PK of SPL84: maximum serum concentration (Cmax) | Predose and 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours postdose, Day 7 and Day 31.
Characterization of PK of SPL84: Time to Cmax (Tmax) | Predose and 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours postdose, Day 7 and Day 31.
Characterization of PK of SPL84: terminal elimination half-life (t1/2) | Predose and 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours postdose, Day 7 and Day 31.
Characterization of PK of SPL84: Area under the curve to the final sample (AUC0-t) | Predose and 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours postdose, Day 7 and Day 31.
Characterization of PK of SPL84: Area under the curve to infinity (AUC0-∞) | Predose and 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours postdose, Day 7 and Day 31.
Characterization of PK of SPL84: Apparent clearance (CL/F) | Predose and 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours postdose, Day 7 and Day 31.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Ein Kerem Hospital Clinical Research Center, Jerusalem, Israel